CLINICAL TRIAL: NCT00364884
Title: Comparison of the Effects Between Keto-/Amino Acid Supplemented Low Protein Diet and Non-Supplemented Low Protein Diet in Patients With Stage Ⅴ Chronic Kidney Disease
Brief Title: Keto-/Amino Acid Supplemented Low Protein Diet in Patients With Chronic Kidney Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 941213
Record Dates: First submitted 2006-08-15; First posted 2006-08-16 (Estimated); Last update posted 2006-08-16 (Estimated); Status verified 2006-08

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

INTERVENTIONS:
Drug: ketoaminoacid

SUMMARY:
Keto-/amino acid supplemented low protein diet can reduce uremic symptoms, improve nutritional status, delay dialysis therapy and enhance health-related quality of life in our patients with stage V CKD in comparison to non-supplemented low protein diet.

DETAILED DESCRIPTION:
Fifty patients will be included into the study. The study comprises 9 visits. The treatment period covers 6 months, preceded by a 2-week screening period and a 1 month run-in period. Patients are required to visit the investigator two times before the start of active treatment.

All patients who are qualified for this study will then be randomised by receiving their medication/introduction of dietary management using the standard simple randomization method.Group I patients will receive keto-/amino acid (Ketosteril) supplemented low protein diet during the active treatment period while Group II patients will receive non-supplemented low protein diet during the same period. The daily dose of keto-/amino acid for each Group I patient is one tablet every 5 kg body weight. The total daily dose will be divided into three times a day.

ELIGIBILITY:
Inclusion Criteria:

* 1. Serum creatinine ≧6 mg/dl at Visit 12. Creatinine clearance < 15 ml/min at Visit 13. Urine output ≧ 1,000 ml/day4. Primary renal disease: chronic glomerulonephritis or non-diabetic stage Ⅴ chronic kidney disease (confirmed by biopsy or clinical presentations/symptoms)5. Bilaterally reduced renal size shown by sonography6. Male or female patients aged 20 - 657. Ability of the patient to understand the basic implications of the study and to follow instructions8. Willingness to participate as indicated by a signed written informed consent

Exclusion Criteria:

* 1. Severe arterial hypertension not responsive to medical therapy, maximum blood pressure values allowed: 180/100 mm Hg 2. Inadequate caloric intake due to extremely severe uremia (vomiting, anorexia, etc) 3. Malnutrition status with serum albumin level less than 3.5 g/dl in recent one month 4. Lack of adherence to dietary prescription 5. Water and sodium retention not responsive to diuretics 6. Clinical relevant severe cardiac disease, hepatic disorders (total bilirubin > 1.5 times the upper limit of normal), malabsorption disorders, diseases requiring steroids or non-steroid anti-inflammatory drugs 7. Severe sodium wasting syndrome that may affect renal function markedly and independently of dietary therapy 8. Concurrent use of nephrotoxic drugs 9. Severe infection with catabolic situation 10. Signs of uremic pericarditis 11. Symptoms of uremic polyneuropathy 12. Disorder of amino acid metabolism 13. Pregnant or nursing women 14. Participation in a clinical trial within the last 2 months 15. Former participation in the present study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2006-08; Study Completion 2007-08

PRIMARY OUTCOMES:
Glomerular filtration rate (GFR) and creatinine clearance (Ccr)

SECONDARY OUTCOMES:
1. Hemodynamics, 2. Biochemistry status, 3. Bone density analysis, 4. Nutritional status, 5. Urinary status, 6. Compliance check, 7. Incidence of Aes8. Health-related quality of life, 9. Economic benefit

CONTACTS AND LOCATIONS:
Overall Officials: Kao Tze-Wah, MD, Master, Principal Investigator — National Taiwan University Hospital